CLINICAL TRIAL: NCT00027768
Title: Randomised Trial of Adjuvant Hepatic Intra-Arterial Iodine-131-Lipiodol Following Curative Resection of Hepatocellular Carcinoma
Brief Title: Radioactive Iodine in Treating Patients Who Have Undergone Surgery for Liver Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Medical Research Council (NMRC), Singapore (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069066; NMRC-AHCC03; EU-20128
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-06

CONDITIONS: Liver Cancer
Keywords: localized resectable adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Chemotherapy, Adjuvant

INTERVENTIONS:
Procedure: adjuvant therapy
Radiation: iodine I 131 ethiodized oil

SUMMARY:
RATIONALE: Radioactive iodine may be effective in reducing the rate of recurrence of liver cancer after surgery to remove the tumor. It is not yet known if radioactive iodine is more effective than no further treatment after surgery.

PURPOSE: Randomized phase III trial to determine the effectiveness of radioactive iodine in treating patients who have undergone surgery for liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of adjuvant hepatic intra-arterial iodine I 131 lipiodol vs observation in terms of rate of recurrence and overall survival of patients with curatively resected hepatocellular carcinoma.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Within 4-6 weeks after prior resection, patients receive adjuvant hepatic intra-arterial iodine I 131 lipiodol once.
* Arm II: After prior resection, patients undergo observation. Patients are followed monthly for 1 year and then every 3 months thereafter.

PROJECTED ACCRUAL: A minimum of 300 patients (150 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary hepatocellular carcinoma (HCC)
* Completely resected disease with clear margins
* No residual disease by postoperative CT scan
* No metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 17 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 1,500/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin less than 2.92 mg/dL
* PT less than 4 seconds over control

Renal:

* Creatinine less than 2.26 mg/dL

Other:

* No contraindication to contrast or radioactive iodine
* No uncontrolled thyrotoxicosis
* No other prior or concurrent malignancy
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* No other prior treatment for HCC

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2001-06

PRIMARY OUTCOMES:
Recurrence-free survival

SECONDARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: London L. Ooi Peng Jin, MD, Study Chair — National Cancer Centre, Singapore
Locations (3):
- Singapore (3):
  - National Cancer Centre - Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore